CLINICAL TRIAL: NCT05971485
Title: Efficacy of Melatonin As an Analgesic in Preterm Neonate
Brief Title: Melatonin As an Analgesic in Preterm Neonate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU MS 496/2022
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-12

CONDITIONS: Preterm Neonate Analgesia
Keywords: Preterm; Analgesia; Melatonin; Oxidative stress
MeSH Terms: conditions — Premature Birth; Agnosia | interventions — Melatonin

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Melatonin group (Experimental): Preterm neonates will receive melatonin 30 minutes before the venous cannula insertion.
  Interventions: Drug: Melatonin 10 mg
- Placebo group (Placebo Comparator): Preterm neonates will receive 2 ml of distilled water as a placebo 30 minutes before venous cannula insertion.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Melatonin 10 mg — Melatonin 10 mg will be used. 5 mg·kg-1 dissolved in 2 ml of distilled water via enteral route in one single dose 30 minutes before the venous cannula insertion
  Arms: Melatonin group
Other: Placebo — The placebo group will receive 2 ml of distilled water as a placebo 30 minutes before venous cannula insertion.
  Arms: Placebo group

SUMMARY:
Melatonin (N-acetyl-5-methoxytryptamine) is a neurohormone secreted by the pineal gland with several important functions, including regulation of the circadian rhythms, antioxidant and anti-inflammatory effects, accumulating evidence revealed that it also plays an important role in pain modulation through multiple mechanisms. The investigators aimed to evaluate the analgesic effect of enteral melatonin given 30 minutes before cannula insertion in preterm neonates by assessing Premature Infant pain Profile score (PIPP) before and 5 minutes after the procedure. Additionally, the study aimed to explore the relationship between procedural pain and oxidative stress, along with the effectiveness of pain management of melatonin by measuring Malondialdehyde (MDA), a well-accepted marker of oxidative stress, 60 minutes after the procedure.

DETAILED DESCRIPTION:
This is a randomized, double-blind, controlled trial

ELIGIBILITY:
Inclusion Criteria:

* Preterm infant
* less than 37 weeks gestational age
* who started enteral feeding.

Exclusion Criteria:

* Multiple congenital anomalies.
* Facial malformation.
* Receiving analgesia or sedation.
* Contraindication of enteral feeding.
* Clinical or laboratory signs of sepsis.
* Infants with high oxygen needs either on invasive or non-invasive mechanical ventilation.

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2022-08-20 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the analgesic effect of melatonin in preterm | 5 minutes starting just before cannula insertion to 5 minutes after the procedure
  Evaluate the analgesic effect of melatonin during venous cannula insertion in preterm neonates by assessing Premature Infant pain Profile score (PIPP) before and 5 minutes after the procedure.
  Premature Infant pain Profile score (PIPP) scale 0-21, with 0-6 reflecting no pain, 6-12 reflecting mild-moderate pain, and above 12 indicating severe pain
Malondialdehyde (MDA), marker of oxidative stress | 60 minutes of the procedure
  Serum Malondialdehyde (MDA), a marker of oxidative stress through measuring serum MDA after 60 minutes of the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine - Ain Shams University, Cairo, Egypt